CLINICAL TRIAL: NCT04170517
Title: Serum Progesterone Levels on the Day of Frozen Embryo Transfer (FET) and Pregnancy Outcomes
Acronym: ProFET
Status: Completed | Type: Observational
Sponsor: CARE Fertility UK (Other)
Responsible Party: Sponsor
Other Study IDs: ProFETStudy
Record Dates: First submitted 2019-11-12; First posted 2019-11-20 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Infertility; Infertility, Female; IVF
MeSH Terms: conditions — Infertility; Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum progesterone will be measured from consenting participants on the day of frozen embryo transfer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measurement of serum progesterone on the day of FET — Measurement of serum progesterone on the day of FET

SUMMARY:
Frozen embryo transfer (FET) cycles have become more common in recent years due to a push towards elective single embryo transfer (SET). While it is known that progesterone supplementation during the luteal phase improves clinical pregnancy rates, there is a paucity of prospective data on the impact of serum progesterone levels on pregnancy outcomes in FET cycles. This multicentre prospective cohort study aims to investigate the association between serum progesterone levels on the day of FET and pregnancy outcomes, and to determine a serum progesterone cut-off value above which clinical pregnancy and live birth are more likely to occur. Women undergoing ART-FET cycles at CARE Fertility clinics in the UK will be recruited and their serum progesterone measured on the day of frozen embryo transfer. Follow-up data will be stored in electronic patient records and analysed to determine whether a low serum progesterone level on the day of FET adversely affects ART outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All women undergoing ART with FET.

Exclusion Criteria:

* None. We aim to study the "every day" patient undergoing FET, and for this we intend to keep the population of the study as unselected as possible.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All women undergoing ART with FET.
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Live birth rate per participant | 18 months
  Birth of a live fetus at 24 or more weeks of gestational age

SECONDARY OUTCOMES:
Miscarriage rate per participant and per pregnancy | 18 months
  Any clinical pregnancy lost before week 12 of gestation per participant (number of events/number of participants, %)
Implantation rates per participant | 18 months
  Number of gestational sacs seen in a 2D transvaginal ultrasound scan divided by the number of embryos transferred per patient (number of events/number of embryos transferred, %)
Biochemical pregnancy rate per participant | 18 months
  Positive pregnancy test following embryo transfer per participant (number of events/number of participants, %)
Clinical pregnancy rate per participant | 18 months
  Presence of at least one gestational sac on ultrasound (number of events/number of participants, %)
Ectopic pregnancy rate per participant | 18 months
  number of events/number of participants, %

CONTACTS AND LOCATIONS:
Overall Officials: Arri Coomarasamy, MBChB MD FRCOG, Principal Investigator — CARE Fertility UK
Locations (1):
- CARE Fertility Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers. Any IPD will be confined to the purposes of the study.

REFERENCES:
- [Derived] Melo P, Wood S, Petsas G, Chung Y, Easter C, Price MJ, Fishel S, Khairy M, Kingsland C, Lowe P, Rajkhowa M, Sephton V, Pandey S, Kazem R, Walker D, Gorodeckaja J, Wilcox M, Gallos I, Tozer A, Coomarasamy A. The effect of frozen embryo transfer regimen on the association between serum progesterone and live birth: a multicentre prospective cohort study (ProFET). Hum Reprod Open. 2022 Nov 28;2022(4):hoac054. doi: 10.1093/hropen/hoac054. eCollection 2022. PMID 36518987